CLINICAL TRIAL: NCT06678529
Title: Effect of Transcranial Direct Current Stimulation on Postoperative Delirium in Elderly Patients Undergoing Hip Fracture Surgery
Brief Title: Effect of Transcranial Direct Current Stimulation on Postoperative Delirium in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hua Zheng, Head of the Anesthesiology Department, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YXLL-2024-191
Record Dates: First submitted 2024-10-18; First posted 2024-11-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Delirium - Postoperative; Hip Fractures (ICD-10 72.01-72.2)
MeSH Terms: conditions — Emergence Delirium; Hip Fractures

STUDY DESIGN:
Intervention Model Description: The tDCS procedure is administered using a transcranial direct current stimulator, with two electrodes placed in physiological saline soaked sponges. The electrodes are secured with a stretchable cap, positioning the anode over the left dorsolateral prefrontal cortex (DLPFC) and the cathode over the right supraorbital area. The active-tDCS group will receive a 15-second ramp up phase at the start, 2 mA of tDCS for 20 minutes and a 15-second ramp down phase at the end. The sham-tDCS group will only receive the 15-second ramp up phase at the beginning and the 15-second ramp down phase at the end of each session, without the continuous 2 mA current for 20 minutes .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants will remain blinded to their group assignment. Surgeons, anesthesiologists, and ward and operating room nurses will also be blinded to the group allocations and intervention protocols. Additionally, personnel involved in outcome assessment, follow-up, data collection, and data processing will remain blinded to both the intervention protocols and group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- active tDCS (Active Comparator): The active-tDCS group will receive a 15-second ramp up phase at the start, 2 mA of tDCS for 20 minutes and a 15-second ramp down phase at the end.
  Interventions: Device: active tDCS
- sham tDCS (Sham Comparator): The sham-tDCS group will only receive the 15-second ramp up phase at the beginning and the 15-second ramp down phase at the end of each session, without the continuous 2 mA current for 20 minutes
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — The active-tDCS group will receive a 15-second ramp up phase at the start, 2 mA of tDCS for 20 minutes and a 15-second ramp down phase at the end.
  Arms: active tDCS
Device: sham tDCS — The sham-tDCS group will only receive the 15-second ramp up phase at the beginning and the 15-second ramp down phase at the end of each session, without the continuous 2 mA current for 20 minutes
  Arms: sham tDCS

SUMMARY:
To evaluate the efficacy of transcranial direct current stimulation (tDCS) in reducing the incidence of postoperative delirium (POD) in elderly patients undergoing hip fracture surgery.

This single-center, double-blind, randomized controlled trial will enroll participants aged 65 years and older, scheduled for elective hip surgery under spinal anesthesia. Participants will be randomly assigned to either the active-tDCS group or the sham-tDCS group. The active-tDCS group will receive two sessions: one pre-surgery and one post-surgery, with electrodes positioned over the left dorsolateral prefrontal cortex and the right supraorbital area. Each session includes 15-second ramp-up phase at the start, 20 minutes simulation with 2 mA current and 15-second ramp-down phase at the end. The sham-tDCS group will receive two sham procedures with no actual current delivered. Functional brain activity will be monitored before and after each session or sham procedure to assess changes in cortical activation and connectivity using functional near-infrared spectroscopy (fNIRS). The primary outcome measure will be the incidence of POD, assessed using the 3-Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM). Secondary outcomes include the severity of delirium, postoperative pain, anxiety, depression, cognitive function, and sleep quality.

DETAILED DESCRIPTION:
1. Screening The trial staff will review orthopedic inpatient registration lists and elective surgery application forms to identify adults aged 65 years and older scheduled for surgical repair of clinically or radiologically diagnosed femoral neck, intertrochanteric, or subtrochanteric hip fractures. Potential participants will be screened for eligibility based on inclusion and exclusion criteria, which will be assessed through medical record reviews and face-to-face interviews.
2. Specific intervention The standard intervention consists of two sessions of tDCS and four sessions of fNIRS. The tDCS sessions will be administered on the day of surgery: the first session will be conducted preoperatively and the second session will take place postoperatively in the PACU. The fNIRS assessments will be performed as part of the monitoring protocol at four designated time points throughout the study.
3. Four fNIRS procedures will be conducted in relation to the tDCS interventions: (1) f1 (pre first tDCS) will be conducted before the first tDCS session; (2) f2 (post first tDCS, pre-surgery) will be conducted after the first tDCS session and before surgery; (3) f3 (post-surgery, before second tDCS) will be conducted after surgery and before the second tDCS session; (4) f4 (post second tDCS) will be conducted after the second tDCS session.

The primary outcome measure will be the incidence of POD, assessed using the 3-Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM). Secondary outcomes include the severity of delirium, postoperative pain, anxiety, depression, cognitive function, and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

(1) aged ≥ 65 years; (2) scheduled for elective hip fracture, including femoral head fractures, femoral neck fractures, intertrochanteric or subtrochanteric fractures, femoral head replacement, total hip arthroplasty, or open or closed reduction; (3) platelet count > 80 × 10⁹/L; (4) ASA classification ≤ Grade III; (5) Mini-Mental State Examination (MMSE) scores ≥ 18 points (13); (6) willingness to participate and sign the informed consent form.

Exclusion Criteria:

(1) severe mental disorders,(e.g,depression or schizophrenia requiring medication treatment); (2) cranial or scalp injuries; (3) history of symptomatic cerebrovascular disease, including stroke, transient ischemic attack; (4) compound injuries, multiple fractures, periprosthetic fractures, and hip joint revisions; (5) drug or alcohol abuse; (6) severe visual or hearing impairments; (7) history of epilepsy or intracranial metal implants; (8) severe cardiovascular disease history and liver dysfunction, or kidney dysfunction; (9) coagulation abnormalities; (10) severe chronic obstructive pulmonary disease; (11) participation in other clinical studies within the past 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | postoperative days 1, 2 and 3
  Delirium will be assessed during the first three postoperative days.The Confusion Assessment Method (CAM) assessment is based on the four key features of delirium: acute onset and fluctuating course, disorganized thinking, inattention, and altered levels of consciousness. Investigators will also consult the medical record or contact a family member, friend, or health care provider who knows the patient well to gather additional information regarding the patient's symptoms.

SECONDARY OUTCOMES:
Subtypes of postoperative delirium. | postoperative days 1, 2 and 3
  Delirium subtypes will be assessed using the Richmond Agitation Sedation Scale (RASS) . Hyperactive delirium is characterized by symptoms ranging from mild restlessness to persistent motor activity and irritability. Conversely, hypoactive delirium is characterized by one or more of the following features: reduced or absent movement, minimal verbal communication despite stimulation, and a lack of responsiveness. Mixed delirium is characterized by rapid fluctuations between the hyperactive and hypoactive states.
pain score | postoperative days 1, 2 and 3
  Pain at rest and during movement will be assessed using the Numeric Rating Scale (NRS) , an 11-point scale where 0 denotes no pain and 10 represents the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zheng, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
Paper case report forms were written by hand

REFERENCES:
- [Derived] Xue LC, Ji HJ, Fan SS, Niu Q, Zhang JY, Fang AL, Wang PZ, Tian SY, Zheng H. Effect of transcranial direct current stimulation on postoperative delirium in elderly patients undergoing hip fracture surgery: study protocol for a randomized controlled trial. Front Med (Lausanne). 2025 May 15;12:1558376. doi: 10.3389/fmed.2025.1558376. eCollection 2025. PMID 40443512